CLINICAL TRIAL: NCT07368478
Title: A Phase Ⅰa/Ⅰb, Open-Label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Preliminary Efficacy of BC2027 in Patients With Advanced Solid Malignancies
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Preliminary Efficacy of BC2027 in Patients With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC2027-102
Record Dates: First submitted 2026-01-12; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Malignancies
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BC2027 treatment group (Experimental): BC2027 is administered via IV infusion, with 2 phases:
  * Phase Ia (dose escalation): 4 levels (0.8/1.2/1.8/2.4 mg/kg); first 3 levels: Q2W (28-day cycle); 4th level: simultaneous exploration of Q2W (28-day cycle) and Q3W (21-day cycle).
  * Phase Ib (dose expansion): 3 GPC3-positive cohorts (NSCLC/HCC/others) treated at Phase Ia's recommended dose.
  Interventions: Drug: BC2027 for Injection

INTERVENTIONS:
Drug: BC2027 for Injection — Drug: BC2027 for Injection (lyophilized powder, 20 mg/vial) Administration: Administered via intravenous (IV) infusion, with dosing and frequency determined according to Phase Ia (dose escalation) and Phase Ib (dose expansion) study design.

SUMMARY:
This is a phase Ia/Ib, open-label, dose escalation and dose expansion study designed to evaluate the safety, tolerability, PK, and preliminary anticancer activity of BC2027 in patients with advanced solid Malignanciesr

DETAILED DESCRIPTION:
This is a phase Ia/Ib, open-label, dose escalation and dose expansion study designed to evaluate the safety, tolerability, PK, and preliminary anticancer activity of BC2027 in patients with advanced solid Malignanciesr.

This study will consist of two parts: Part 1, a dose escalation part (Phase Ia) and Part 2, a dose expansion part (Phase Ib). Both parts will include a screening period (within 28 days prior to dosing), a treatment period (Q2W(28-day cycle), Q3W(21-day cycle)), a safety follow-up period (45 days (±5 days) after last dose), and a survival follow-up period (every 12 weeks until death)

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Be at least 18 years old.
3. Have an Eastern Cooperative Group (ECOG) performance status (PS) of 0 or 1.
4. Have a life-expectancy of at least 3 months based on the Investigator's assessment.
5. Patients with advanced solid tumors confirmed by histology or cytology, who have failed standard therapy, have no available standard therapy, or are intolerant to standard therapy.
6. Phase 1a (dose escalation, Part 1)

   a. Have an advanced solid malignancy confirmed by histologic or cytologic examination that is known to express GPC3 including, but not limited to, HCC, NSCLC (particularly squamous cell NSCLC), sarcoma (undifferentiated), ovarian clear cell adenocarcinoma (OCCC), esophageal squamous cell carcinoma (ESCC).
7. Must provide either a previously archived tumor tissue sample or a fresh core or excisional biopsy from a site that was not irradiated. There must be at least 3-5 unstained sections. A formalin-fixed, paraffin-embedded (FFPE) tissue block is preferred to slides, and fresh biopsies are preferred over archival tissue. If archival tissue cannot be provided and a fresh biopsy cannot be obtained in Part 1, an exemption may be provided by the Sponsor.
8. Must have adequate organ function within 7 days prior to the start of study treatment as defined below:

   Hematological* ANC ≥1,500/μL or ≥1.5×109/L Platelets ≥100,000/μL or ≥100×109/L (For HCC patients, PLTs ≥75×109/L) Hemoglobin ≥9.0 g/dL Kidney Function Creatinine clearance (CrCl)** ≥50 mL/min Liver Function Total Bilirubin (TBIL) ≤1.5×ULN, or direct bilirubin ≤ULN (patients with total bilirubin level >1.5×ULN).

   AST (SGOT) and ALT (SGPT) ≤2.5×ULN (≤5×ULN in patients with liver metastases) Coagulation International Normalized Ratio (INR), Prothrombin Time (PT), and activated partial thromboplastin time (aPTT) :INR≤1.5; PT and aPTT ≤1.5×ULN or within a therapeutic range if on an anticoagulant.

   * Blood transfusion or growth factor support is not allowed within 14 days prior to blood sampling.

   ** CrCl should be calculated according to institutional standards.
9. Must have at least one measurable tumor lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (In the dose escalation part of the study (Part 1), patients without measurable lesions may be enrolled if they have evaluable disease and are approved by the sponsor). Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
10. Must agree to use highly effective contraceptive measures if patient is a man or woman of childbearing potential. Highly effective contraceptive measures include measures like hormonal contraceptives, intrauterine devices, vasectomy, or tubal ligation, and others (Section 5.3), from the time of signing the informed consent until 6 months after the last dose of the study drug. Women of childbearing potential (WCBP) must have a negative blood or urine pregnancy test within 7 days prior to the first dose of study drug. Female patients with surgically sterile or are postmenopausal for at least 12 months without an alternative medical cause are also allowed.

Additional Inclusion Criteria for Part 2

In addition to fulfilling the inclusion for Part 1, patients enrolling in cohorts in Part 2/Phase Ib must have:

1. Cohort 1 (NSCLC Cohort)

   1. Positive expression of GPC3 confirmed by immunohistochemistry (IHC) assay, or with existing prior IHC test report documenting GPC3 positivity.
   2. Patients with non-small cell lung cancer (NSCLC) who have failed no more than 3 prior lines of systemic antineoplastic therapy.
2. Cohort 2 (HCC Cohort)

   1. IHC evidence of GPC3 expression on archival tumor or a fresh biopsy unless biopsy is not feasible or safe and with approval of the Sponsor.
   2. The subject has received treatment with 1 prior regimen in the first line advanced setting consisting of an appropriate monoclonal antibody (mAb) targeting PD-1 or PD-L1 with an appropriate mAb targeting CTLA-4 and/or an appropriate tyrosine kinase inhibitor (TKI) or mAb targeting vascular endothelial growth factor (VEGF, e.g., bevacizumab). The subject must have progressed, demonstrated intolerance, or refused such treatment. If a subject had refused treatment, the reasons for such must be documented in the records and case report form (CRF).
   3. The patient must have Barcelona Clinic Liver Cancer (BCLC) stage B or C HCC (See Appendix 1), not amenable to locoregional therapy or refractory to locoregional therapy likely to result in reasonable clinical benefit, and not amenable to a curative treatment approach.
   4. The subject has a Child-Pugh A score (See Appendix 2) within 7 days of study drug treatment.
3. Cohort 3 (Advanced GPC3 expressing solid cancer).

   1. GPC3 positivity confirmed by IHC assay, or documented in prior IHC reports.
   2. Patients excluding Cohort 1 and Cohort 2 with failure of ≤ 2 prior lines of systemic antineoplastic therapy.

Exclusion Criteria:

Patients who meet any of the exclusion criteria must not be enrolled in the study.

1. Prior treatment with GPC3-targeted ADC.
2. Prior treatment with systemic anticancer treatment, including investigational agents, within a period that is less than five half-lives or 2 weeks before the start of treatment, whichever is shorter.
3. Known hypersensitivity or delayed hypersensitivity reactions to the same class and/or any component of BC2027.
4. Treatment with strong CYP3A4 inhibitors or inducers, and P-gp inhibitors within 14 days or 5 half-lives whichever is shorter, before the first dose.
5. For patients with advanced NSCLC:

   a. Positive for driver oncogenes: including EGFR mutation, ALK gene fusion, ROS1 gene fusion, KRAS-G12C mutation, c-MET (exon 14 skipping, MET amplification and overexpression), HER2 mutation, RET gene fusion, etc.

   For HCC patients:
   1. Received local hepatic therapy including, but not limited to, surgery, radiotherapy, hepatic arterial embolization (TAE), hepatic arterial chemoembolization (TACE), hepatic arterial perfusion, radiofrequency ablation, cryoablation, or percutaneous ethanol injection) within 4 weeks prior to initiation of the study drug.
   2. History of hepatic encephalopathy within past 12 months or requirement for medications to prevent or control encephalopathy (eg, no lactulose, rifaximin, etc if used for purposes of hepatic encephalopathy)
   3. The patient has main portal vein thrombosis ((i.e. thrombosis in the main trunk of the portal vein, with or without blood flow) on baseline imaging.)
   4. Documented gastrointestinal bleeding within past 6 months or at high risk of gastrointestinal bleeding per investigator's clinical judgement, due to esophageal varices, active gastric or duodenal ulcers.
6. Active and severe viral infections meeting the following criteria:

   1. Known HIV seropositivity.
   2. Known active hepatitis B (Screening for hepatitis B is not required for non-HCC patients):

      * For HCC patients: HBV DNA > 2000 IU/mL. (For patients with positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV DNA (≥10 IU/mL)], patients with the following conditions may be enrolled: patients who have received antiviral therapy and had sufficient suppression of viral replication before enrollment (HBV DNA ≤ 2000 IU/ml), and patients must continue to receive antiviral therapy during the study and for 6 months after the last dose.)
      * For other solid malignancies patients: HBsAg positive and HBV-DNA titer > 500 IU/mL or > 2500 copies/mL.
   3. Known active hepatitis C :

      * For HCC patients: Co-infection of HBV and HCV. (The following conditions are allowed for inclusion: positive HCV RNA test or positive HCV antibody, and patients complying with local medical practice for treatment.)
7. Severe immunodeficiency requiring systemic corticosteroid therapy at a prednisone-equivalent dose (>10 mg/day), or any other systemic immunosuppressive therapy, unless approved by the sponsor.
8. A history of allogeneic tissue or solid organ transplantation.
9. A history of radiation pneumonitis, or receipt of radiotherapy within 2 weeks prior to the initiation of study treatment.

   Note: Patients must have recovered from radiation-related toxicities and must not be receiving corticosteroid treatment. A 1-week washout period is permitted for palliative radiotherapy (≤ 2 weeks of radiotherapy) for non-central nervous system (non-CNS) diseases.
10. Unstable central nervous system (CNS) metastases and/or carcinomatous meningitis. For patients with previously treated brain metastases who have achieved radiological stability (i.e., no evidence of disease progression on repeated imaging examinations for at least 4 weeks, as documented in imaging obtained during screening; and no requirement for corticosteroid treatment for at least 14 days prior to the first dose), routine brain imaging is not required during screening.
11. Uncontrolled pleural effusion, ascites, or pericardial effusion at the time of screening.
12. A history of interstitial lung disease (ILD) or drug-related interstitial lung disease, or any evidence of clinically active interstitial lung disease.
13. Clinically significant cardiovascular disease, including but not limited to:

    * Congestive heart failure (CHF) of New York Heart Association (NYHA) functional class III or higher, or left ventricular ejection fraction (LVEF) < 50%.
    * Unstable angina pectoris or myocardial infarction occurring within 6 months prior to enrollment.
    * Severe cardiac arrhythmias, including but not limited to complete left bundle branch block, atrioventricular block of second degree or higher, and ventricular tachycardia (including frequent ventricular premature beats).
    * Clinically uncontrolled hypertension, defined as systolic blood pressure (SBP) ≥ 160 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg despite anti-hypertensive medication use.
14. Clinically significant electrocardiogram (ECG) abnormalities, including any of the following:

    * Markedly prolonged QT/QTc interval on screening ECG (i.e., repeated measurements demonstrating a QTc interval > 470 ms) (QTcF calculated based on the Fridericia formula).
    * A history of risk factors for torsades de pointes, such as congestive heart failure, hypokalemia, family history of long QT syndrome, and other risk factors.
15. Grade ≥ 2 peripheral neurotoxicity or neuropathy, and other toxicities caused by prior anti-tumor therapy that have not resolved to Grade ≤ 1 (per CTCAE Version 5.0). Exceptions include alopecia, skin hyperpigmentation, other events deemed tolerable by the investigator, or specific-grade toxicities specified in the inclusion/exclusion criteria of this study.
16. Patients with active or chronic corneal disease, other active ophthalmic diseases requiring continuous treatment, or any clinically significant corneal disease that prevents adequate monitoring for drug-induced keratopathy.
17. Active infections requiring systemic anti-infective therapy.
18. Poor patient compliance, or unwillingness or inability to follow the procedures specified in the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Dose limiting toxicities (DLT) will be assessed At the end of Cycle 1 (each cycle is 28 or 21 days).
  The incidence of dose-limiting toxicity (DLT) at different doses of BC2027 in patients with advanced solid malignancies
The safety and tolerability | Through study completion, an average of 2 years.
  To assess the safety and tolerability of BC2027 in patients with advanced solid malignancies
Preliminary antitumor activity | Through study completion, an average of 2 years.
  To assess the preliminary antitumor activity of BC2027 in patients with advanced solid malignancies

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai, China, China